CLINICAL TRIAL: NCT07246096
Title: Exploratory Clinical Study on the Safety and Efficacy of Anti-CD19/BCMA Universal CAR-T Cell Injection for the Treatment of Relapsed/Refractory Autoimmune Diseases
Brief Title: Exploratory Clinical Study on the Safety and Efficacy of Anti- CD19/BCMA U CAR-T Cell Injection for the Treatment of Relapsed/Refractory Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Rui Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2025-363
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Autoimmune Diseases; Systemic Lupus Erythematosus; Systemic Sclerosis; Primary Sjögren Syndrome; Rheumatoid Arthritis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis
MeSH Terms: conditions — Autoimmune Diseases; Lupus Erythematosus, Systemic; Scleroderma, Systemic; Arthritis, Rheumatoid; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN3601 (Experimental)
  Interventions: Biological: anti-CD19/BCMA U CAR T cells

INTERVENTIONS:
Biological: anti-CD19/BCMA U CAR T cells — Patients will receive Fludarabine and Cyclophosphamide on day-5, -4, and -3. Multiple doses of anti-CD19/BCMA CAR T cells (KN3601) will infused using dose-escalation strategy.

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety and effectiveness of anti-CD19/BCMA U CAR T cells in patients with autoimmune diseases.

60 patients are planned to be enrolled in the dose-escalation trial.

ELIGIBILITY:
Common inclusion criteria:

1. Age: ≥ 18 years old and ≤ 70 years old, male or female;
2. The functions of critical organs meet the following requirements:

a )Neutrophil count ≥ 1 x 10^9/L, Hemoglobin ≥60g/L; b) Liver function: ALT ≤ 3 x ULN,AST≤3 x ULN, TBIL≤1.5 x ULN; c) Coagulation function: International standardized ratio (INR) ≤1.5x ULN, prothrombin time (PT) ≤1.5 x ULN; d) Cardiac function: good hemodynamic stability, left ventricular ejection fraction (LVEF) ≥50%; 3. Female subjects of childbearing potential and male subjects whose partner is a female of childbearing potential are required to use medically approved contraception or abstain from sex for at least 6 months during and at least 6 months after the end of the study treatment period; female subjects of childbearing potential have had a negativeserum HCG test within 7 days prior to study enrollment and are not lactating; 4. Voluntarily participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Specific inclusion criteria:

Relapsed/Refractory Systemic lupus erythematosus

1. Subject have previous diagnosis of systemic lupus erythematosus (SLE) (according to the 1997 American College of Rheumatology revised SLE classification criteria, the 2012 Systemic Lupus International Collaborating Clinics classification criteria, or the 2019 European League Against Rheumatism/American College of Rheumatology joint classification criteria);
2. Subjects had a modified SLEDAI-2K score of ≥8 at screening;
3. Subject has ≥ 1 organ system with BILAG-2004 Class A mobility score or ≥ 2 organ systems with BILAG-2004 Class B mobility score at screening;
4. Based on the results of the central laboratory tests at screening, the subject meets one of the following: a. ANA by immunofluorescence ≥ 1:80 b. Anti-dsDNA antibodies above the normal level c. Anti-Smith antibodies above the normal level.

Relapsed/Refractory Systemic Sclerosis

1. Meets 2013 ACR classification criteria for systemic sclerosis;
2. If combined with interstitial pneumonia, interstitial changes suggestive of ground-glass exudates on chest HRCT and FVC or DLCO <70% predictive value on pulmonary function tests;
3. Ineffective conventional treatment or relapse of disease activity after remission. Definition of routine treatment: Use of glucocorticoids (above 1mg/Kg/d) and cyclophosphamide, as well as any of the following immunomodulatory drugs for more than 6 months: antimalarials,
4. methotrexate, leflunomide, cyclophosphamide, azathioprine, mertiomate, tacrolimus, cyclosporine, and biologics, including rituximab, belimumab and tetracycline;
5. Definition of progressiveness; 1) Definition of cutaneous progression: increase in mRSS >10%; 2) Definition of lung disease progression: 10% decrease in FVC or 5% decrease in FVC with 15% decrease in DLCO (OMERACT progression).

Relapsed/Refractory Primary Sjögren's Syndrome

1. Meets 2002 AECG criteria or 2016 ACR/EULAR classification criteria for primary dry syndrome (pSS);
2. Definition of disease activity: investigator-assessed disease ESSDAI score of 5 or higher;
3. Ineffective conventional treatment or relapse of disease activity after remission. Definition of routine treatment: Use of glucocorticoids (above 1mg/Kg/d) and cyclophosphamide, as well as any of the following immunomodulatory drugs for more than 6 months: antimalarials, methotrexate, leflunomide, cyclophosphamide, azathioprine, mertiomate, tacrolimus, cyclosporine, and biologics, including rituximab, belimumab and tetracycline.

Relapsed/Refractory rheumatoid arthritis

1. Meets the diagnostic criteria of the 2010 ACR/EULAR classification. Diagnosis of moderately or severely active rheumatoid arthritis with a previous diagnosis of rheumatoid arthritis ≥ 6 months;
2. A swollen joint count of ≥ 6 (based on 66 joint counts) and a tender joint count of ≥ 6 (based on 68 joint counts) during the Screening Period;
3. C-reactive protein (CRP) ≥ 10 mg/L or erythrocyte sedimentation rate (ESR) ≥ 28 mm/h during the Screening Period;
4. EULAR definition of refractory rheumatoid arthritis:

1） Failure of treatment according to EULAR recommended guidelines and failure of treatment with ≥2 b/tsDMARDs despite failure of treatment with csDMARDs. (i) unless treatment with bDMARDs/tsDMARDs is limited due to socioeconomic factors; and (ii) if treatment with csDMARDs is contraindicated, then failure of treatment with ≥2 b/tsDMARDs of different mechanisms also fulfills the condition); 2） Symptom management of RA is considered problematic by both the patient and the physician; 3） Signs suggestive of active or progressive disease if at least 1 of the following 5 items is met (Meeting all three of the below criteria can be diagnosed as rheumatoid arthritis): i. At least moderate disease activity (DAS28-ESR >3.2 or CDAI>10); ii. Signs and/or symptoms suggestive of active disease; iii. Inability to reduce glucocorticoids to less than 7.5 mg/dayprednisone or equivalent; iv. Rapid imaging progression (1-year increase of ≥5 points in vander Heijde modified Sharp score); v. Decreased quality of life due to RA, although RA is well controlled.

Relapsed/refractory anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis

1. Meets 2022 ACR/EULAR diagnostic criteria for ANCA vasculitis, including microscopic polyangiitis, granulomatous polyangiitis, eosinophilic granulomatous polyangiitis;
2. Positive ANCA related antibodies (MPO-ANCA or PR3-ANCA positive);
3. The Birmingham Vasculitis Activity Scale (BVAS) is ≥ 15 points (a total score of 63 points), indicating the activity of the vasculitis condition;
4. Glomerular filtration rate (eGFR, CKD-EPI formula) ≥15 ml/min/1.73 m2 during the screening period.

Exclusion Criteria:

Subjects who meet any of the following common exclusion criteria or disease-specific exclusion criteria will not be eligible for this study.

Common exclusion Criteria:

1. Subjects with known severe allergic reactions, hypersensitivity, contraindication to any medications during the trial (cyclophosphamide, fludarabine, tozumabs), or subjects with a history of severe allergic reactions;
2. Existence or suspicion of uncontrollable or treatable fungal, bacterial, viral or other infections;
3. Subjects with central nervous system disorders caused by ADs or not caused by ADs (including epilepsy, psychiatric disorders, organic encephalopathy syndromes, cerebrovascular accidents, encephalitis, central nervous system vasculitis);
4. Subjects s with relatively serious heart diseases, such as angina pectoris, myocardial infarction, heart failure, and arrhythmia;
5. Subjects with congenital immunoglobulin deficiency;
6. Subjects with malignant tumors (except for non-melanoma skin cancer and in situ cervical, bladder, and breast cancers that have been disease free for more than 5 years);
7. Subjects with end-stage renal failure;
8. Subjects with positive hepatitis B surface antigen (HBsAg) or hepatitis,B core antibody (HBcAb) and HBV DNA titer in peripheral blood higher than the upper limit of detection; Patients with positive hepatitis C virus (HCV) antibodies and positive peripheral blood HCV RNA; People who are positive for human immunodeficiency virus (HIV) antibodies; Those who have tested positive for syphilis;
9. Subjects with mental illness and severe cognitive impairment;
10. Subjects who have received other clinical trial treatment within 6 months;
11. Pregnant or intending to conceive women;
12. Subjects with hypertension or diabetes that cannot be controlled by medication;
13. In the opinion of the investigator, there are other reasons that prevent some subjects from being included in this study.

Specific exclusion Criteria:

Relapsed/Refractory Systemic lupus erythematosus

1. Except for SLE, any clinically significant history of cardiac, endocrine, blood, liver, immune, metabolic, urinary, pulmonary, neurological, skin, psychiatric, or renal disorders, or other major diseases that may interfere with the administration of KN3601 (as determined by the investigator);
2. Except for SLE, any active skin disease that could interfere with the research evaluation of SLE including but not limited to psoriasis, dermatomyositis, systemic sclerosis, non-SLE cutaneous lupus manifestations (such as cutaneous vasculopathy, periungual capillary dilation, fingertip sclerosis, rheumatoid nodules, erythema multiforme, leg ulcers) or drug-induced lupus.

Relapsed/Refractory Primary Sjögren's Syndrome

1. SSc-like disease caused by environmental, ingestion, or injection factors, accompanied by other autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, polymyositis, etc.).

Relapsed/Refractory dry syndrome

1. Combined cirrhosis of the liver;
2. Combination of aplastic anemia (AA), myelodysplastic syndrome (MDS), or other myeloproliferative disease (MPD).

Relapsed/Refractory rheumatoid arthritis

1. Functional status of rheumatoid arthritis graded at level 4 according to ACR.

Relapsed/refractory ANCA-associated vasculitis

1. Estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m2;
2. If the patient has alveolar hemorrhage invasive lung ventilation is required, estimated to last longer than the screening period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2027-07-20 (Estimated); Study Completion 2028-07-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicity (DLT) | up to 52 weeks after infusion
  To characterize the safety of anti-CD19/BCMA U CAR T Cells (KN3601) for patients with Relapsed/Refractory autoimmune diseases
Incidence of Treatment Emergent Adverse Events (TEAEs) | up to 52 weeks after infusion
  To characterize the safety of anti-CD19/BCMA U CAR T Cells (KN3601) for patients with Relapsed/Refractory autoimmune diseases

SECONDARY OUTCOMES:
The overall response rate (ORR) | up to 52 weeks after infusion
  To characterize the efficacy of anti-CD19/BCMA U CAR T Cells (KN3601) for patients with Relapsed/Refractory autoimmune diseases
Disease control rate (DCR) | up to 52 weeks after infusion
  To characterize the efficacy of anti-CD19/BCMA U CAR T Cells (KN3601) for patients with Relapsed/Refractory autoimmune diseases
B cell depletion rate | up to 52 weeks after infusion
  To characterize the efficacy of anti-CD19/BCMA U CAR T Cells (KN3601) for patients with Relapsed/Refractory autoimmune diseases
B cell reconstitution | up to 52 weeks after infusion
  B cell subsets in peripheral blood measured by flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China